CLINICAL TRIAL: NCT00149149
Title: Use of Zinc Carnosine on Intestinal Permeability in Healthy Volunteers Taking Non-steroidal Anti-inflammatory Drugs (NSAIDs)
Brief Title: Effect of Zinc Carnosine on Intestinal Permeability in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wexham GI Trust (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 05/Q0408/19
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: Reduction in NSAID related gut damage
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Intervention Model Description: Zinc carnosine or placebo for 7 days with 5 days of indomethacin from days 2-7. It was a cross over protocol with 2 week washout inbetween.

ARMS (2):
- Indomethacin treated volunteers (Experimental): 5d of indomethacin treatment (50 mg t.i.d) with ZnC (37.5 mg b.i.d) coadministration.
  Interventions: Other: Zinc Carnosine coadministered with Indomethacin
- Placebo treated volunteers (Placebo Comparator): 5 days of indomethacin treatment (50 mg t.i.d) with placebo coadministration.
  Interventions: Other: Placebo coadministered with Indomethacin

INTERVENTIONS:
Other: Zinc Carnosine coadministered with Indomethacin
  Arms: Indomethacin treated volunteers
Other: Placebo coadministered with Indomethacin
  Arms: Placebo treated volunteers

SUMMARY:
Zinc carnosine is a food supplement which is available in the health food shops. The investigators wish to see if it can reduce intestinal swelling in people who take non-steroidal anti-inflammatory (anti-swelling) drugs (NSAIDs: non-steroidal antiinflammatory drug.).

DETAILED DESCRIPTION:
The study was about exploring the influence of zinc carnosine (ZnC) on changes in small bowel permeability caused by indomethacin.

Healthy volunteers (n = 10) participated in this double-blind randomised controlled crossover protocol. Each arm comprised two baseline urine collections, followed by a third at the end of that study period. In each arm, volunteers took ZnC (37.5 mg twice daily, orally) or placebo for 7 days, with indomethacin for the final 5 days.

Results were expressed as lactulose:rhamnose (L:R) ratios and mean values for each stage were therefore estimated: when taking placebo, volunteers had a threefold increase in L:R ratios in response to indomethacin administration (p,0.01), whereas no increase was seen if ZnC was also being taken.

All 10 participants completed the study without protocol violations. Two of ten participants developed mild nondescript upper abdominal discomfort while taking the indomethacin (control) arm, but completed the course. None reported symptoms during the ZnC (plus indomethacin) arm, and no side effects due to ingestion of ZnC were reported.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years

Exclusion Criteria:

* Conditions known to alter intestinal permeability, eg previous bowel surgery, celiac disease
* Conditions where NSAIDs are contraindicated, eg asthma, renal failure, heart failure
* Diabetes
* Any other serious illness

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2006-05-18 (Actual); Study Completion 2006-05-18 (Actual)

PRIMARY OUTCOMES:
Lactulose:rhamnose ratio - Arm1 (Urine) | day 5
  Lactulose:rhamnose urine ratio in zinc carnosine/indomethacin coadministered patients
Lactulose:rhamnose ratio - Arm2 (Urine) | day 5
  Lactulose:rhamnose urine ratio in placebo/indomethacin coadministered patients

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Playford, MD, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College, London, United Kingdom

REFERENCES:
- [Result] Mahmood A, FitzGerald AJ, Marchbank T, Ntatsaki E, Murray D, Ghosh S, Playford RJ. Zinc carnosine, a health food supplement that stabilises small bowel integrity and stimulates gut repair processes. Gut. 2007 Feb;56(2):168-75. doi: 10.1136/gut.2006.099929. Epub 2006 Jun 15. PMID 16777920
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/16777920/